CLINICAL TRIAL: NCT04184570
Title: Audit of International Intraoperative Hemotherapy and Blood Loss Documentation
Status: Completed | Type: Observational
Sponsor: Dr. Florian Piekarski (Other)
Responsible Party: Sponsor-Investigator, Dr. Florian Piekarski, Principal Investigator, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: KGU_FP_2019_xCA2
Record Dates: First submitted 2019-11-23; First posted 2019-12-03 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Patient Safety; Patient Blood Management
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Trial — Observational Trial

SUMMARY:
The investigator hypotheses anesthetic records do not contain detailed information on hemotherapy and blood loss estimation. Therefore anesthetic records will be collected from different institutions and analyzed for items concerning hemotherapy contained.

DETAILED DESCRIPTION:
The anaesthetic record is the primary way anesthetists document and communicate information regarding hemotherapy. Records vary in content and design. Several organizations published recommendations, but perioperative hemotherapy is not sufficiently detailed for the purpose.

Anesthetic records will be analyzed for 20 defined hemotherapy and monitoring items by two independent investigators. Disagreements will be resolved by a the principle investigator.

ELIGIBILITY:
Inclusion Criteria:

* Anesthetic records

Exclusion Criteria:

* Incomplete records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: International anesthetic records
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Contained items in anesthetic records | 11/01/2019 - 12/01/2019
  The main outcome measure are hemotherapy-items in anesthetic records

CONTACTS AND LOCATIONS:
Overall Officials: Florian Piekarski, Dr. med., Principal Investigator — Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Frankfurt, Goethe University, Frankfurt, Germany.
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital Frankfurt, Goethe University, Frankfurt, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No